CLINICAL TRIAL: NCT04247490
Title: Multicentric Study on the Long-term Follow-up of Autoimmune Hepatitis in the Pediatric Patients
Brief Title: Autoimmune Hepatitis in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Giuseppe Maggiore, Full Professor, University Hospital of Ferrara
Other Study IDs: 637/2019/Oss/AOUFe
Record Dates: First submitted 2020-01-20; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune hepatitis; incidence; prevalence; immunosuppressive treatmen; liver transplantation
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric AIH: Patients diagnosed with hepatitis type 1 and type 2 formulated between the ages of 0 and 18.
  Interventions: Diagnostic Test: pediatric AIH

INTERVENTIONS:
Diagnostic Test: pediatric AIH — pediatric patients with clinical, laboratory (transaminase and IgG increase), instrumental (ultrasound, liver biopsy) characteristics

SUMMARY:
Autoimmune hepatitis (AIH) is an immune-mediated and inflammatory liver disorder. It is currently divided into types 1 and 2, differentiated and defined by the presence of specific autoantibodies. The objectives are to describe the prevalence and incidence of type 1 and 2 autoimmune hepatitis and to analyze the clinics, biochemical and histopathological profiles at diagnosis and follow-up, initial therapy, response to therapy and long-term follow-up in three Italian centers of patients with type 1 and type 2 AIH.

DETAILED DESCRIPTION:
Background: Autoimmune hepatitis (AIH) is an immune-mediated and inflammatory liver disorder with typical onset in pediatric age. It is currently divided into types 1 and 2, differentiated and defined by the presence of specific autoantibodies. AIH type 1 (AIH-1) is characterised by smooth muscle and/or antinuclear autoantibodies (SMA/ANA) while anti-liver kidney microsomal (anti-LKM) or liver cytosol type 1 (anti-LC1) identified AIH type 2 (AIH-2). The conventional treatment is based on corticosteroids and azathioprine as first line therapy. The optimal duration is not clear definied, however it should be extended for at least five years due to the frequent relapses.

Aims of the study: The primary objective is to describe the prevalence and incidence of type 1 and 2 autoimmune hepatitis on a selected italian pediatric population. Secondary objectives are to analyze the clinical, biochemical and histopathological profiles at diagnosis and follow-up, type of treatment received, response to therapy and long-term follow-up.

Methods: The investigators conducted a retrospective and prospective cohort study on patients aged ≤ 18 years who the diagnosis of AIH 1 and 2 between 01/01/1989 and 31/12/2019 and were followed in three Italian pediatric centers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 18 years at the time of diagnosis
* Diagnosis of autoimmune hepatitis type 1 or 2 according to the Mieli-Vergani score: a pre-treatment score> 15 or post-treatment> 17 indicates a definite diagnosis of Autoimmune Hepatitis; a pre-treatment score between 10 and 15 or post-treatment between 12 and 17 indicates a probable diagnosis.

Exclusion Criteria:

* Age> 18 years at the time of diagnosis
* Presence of other causes of liver disease
* Presence of overlap syndrome (hepatito-cholangitis)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population is represented by all the patients who presented the onset of Autoimmune hepatitis type 1 and type 2 from 01/01/1989 to 31/12/2019 and were followed at the Pediatric Hepatology Centers of Ferrara (Hospital Saint Anna of Cona), Naples (Federico II University Hospital) and Palermo (Mediterranean Institute for Transplants and Highly Specialized Therapies).
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence and incidence | from 01/01/1989 to 31/12/2019
  The primary objective was to calculate the proportion of AIH type 1 and 2 patients present in the Italian pediatric population at a given time (prevalence) and the proportion of new AIH type 1 and 2 patients in the Italian pediatric population (0-18 years) in a given period of time (incidence).

SECONDARY OUTCOMES:
Characteristics of AIH in pediatric patients | from 01/01/1989 to 31/12/2019
  Describe the baseline characteristics (age of onset, clinical-laboratory, radiological and histological characteristics), the response to therapy (medical and / or the possible use of liver transplantation) and the follow-up of patients with autoimmune hepatitis type 1 and 2.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Cona, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jimenez-Rivera C, Ling SC, Ahmed N, Yap J, Aglipay M, Barrowman N, Graitson S, Critch J, Rashid M, Ng VL, Roberts EA, Brill H, Dowhaniuk JK, Bruce G, Bax K, Deneau M, Guttman OR, Schreiber RA, Martin S, Alvarez F. Incidence and Characteristics of Autoimmune Hepatitis. Pediatrics. 2015 Nov;136(5):e1237-48. doi: 10.1542/peds.2015-0578. Epub 2015 Oct 19. PMID 26482664
- [Result] Verma S, Torbenson M, Thuluvath PJ. The impact of ethnicity on the natural history of autoimmune hepatitis. Hepatology. 2007 Dec;46(6):1828-35. doi: 10.1002/hep.21884. PMID 17705297
- [Result] Nastasio S, Sciveres M, Matarazzo L, Maggiore G. Old and New Treatments for Pediatric Autoimmune Hepatitis. Curr Pediatr Rev. 2018;14(3):187-195. doi: 10.2174/1573396314666180516130314. PMID 29766815
- [Result] Maggiore G, Porta G, Bernard O, Hadchouel M, Alvarez F, Homberg JC, Alagille D. Autoimmune hepatitis with initial presentation as acute hepatic failure in young children. J Pediatr. 1990 Feb;116(2):280-2. doi: 10.1016/s0022-3476(05)82892-6. No abstract available. PMID 2299503
- [Result] Alvarez F, Berg PA, Bianchi FB, Bianchi L, Burroughs AK, Cancado EL, Chapman RW, Cooksley WG, Czaja AJ, Desmet VJ, Donaldson PT, Eddleston AL, Fainboim L, Heathcote J, Homberg JC, Hoofnagle JH, Kakumu S, Krawitt EL, Mackay IR, MacSween RN, Maddrey WC, Manns MP, McFarlane IG, Meyer zum Buschenfelde KH, Zeniya M, et al. International Autoimmune Hepatitis Group Report: review of criteria for diagnosis of autoimmune hepatitis. J Hepatol. 1999 Nov;31(5):929-38. doi: 10.1016/s0168-8278(99)80297-9. No abstract available. PMID 10580593
- [Result] Mieli-Vergani G, Vergani D, Baumann U, Czubkowski P, Debray D, Dezsofi A, Fischler B, Gupte G, Hierro L, Indolfi G, Jahnel J, Smets F, Verkade HJ, Hadzic N. Diagnosis and Management of Pediatric Autoimmune Liver Disease: ESPGHAN Hepatology Committee Position Statement. J Pediatr Gastroenterol Nutr. 2018 Feb;66(2):345-360. doi: 10.1097/MPG.0000000000001801. PMID 29356770